CLINICAL TRIAL: NCT02201927
Title: Galvanic Vestibular Stimulation : Role in the Improvement of Egocentric Frame in Patient With Right Parietal Lobe Lesions
Brief Title: Stimulation Galvanique Vestibulaire
Acronym: GVS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of performance
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Collaborators: University of Versailles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2013-A01243-42/1
Record Dates: First submitted 2014-07-22; First posted 2014-07-28 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Hypertensive Hemorrhage of Right Parietal Lobe
Keywords: galvanic vestibular stimulation; right parietal lobe lesion; egocentric space

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- patient with right parietal lobe lesion (Experimental): Patient with right parietal lobe lesion
  Interventions: Device: galvanic vestibular stimulation
- patient stroke (Experimental): patient with cerebral vascular accident
  Interventions: Device: galvanic vestibular stimulation
- healthy volunteers (Experimental): healthy volunteers
  Interventions: Device: galvanic vestibular stimulation

INTERVENTIONS:
Device: galvanic vestibular stimulation
  Other Names: deviation from target score with and without galvanic vestibular stimulation

SUMMARY:
Right posterior parietal cortex is involved in spatial cognition. Blindfolded patients suffering right posterior parietal lesions fail to update their own position after a body rotation. Right cathodal galvanic vestibular stimulation activates right posterior parietal cortex and reduces symptoms of spatial neglect, another disability frequently encountered after right posterior parietal lesion. The aims of this study are to confirm posterior parietal involvement in automatic updating of body-centered spatial relationships and to evaluate therapeutic effects of galvanic vestibular stimulation. Performances of three groups of adults are compared before and during galvanic vestibular stimulation on a pointing task: a healthy control group, a brain-injured control group with stroke lesions sparing right posterior parietal cortex and a group of stroke patients with right posterior parietal lesions.

ELIGIBILITY:
Inclusion Criteria:

* patient with right posterieur parietal lobe lesion
* patient with cerebral vascular stroke
* healthy volonteers Age greater than or equal to 18 written informed consent

Exclusion Criteria:

* patient's refusal to participate to the study
* inability to cooperate
* cognitive trouble
* epilepsy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
deviation from target score | 30 min
  difference in degree between the actual and target score

SECONDARY OUTCOMES:
deviation from target "straight ahead" | 30min
  difference in degree between the actual straight ahead and target score
deviation rightward line bisection | 30min
  percentage difference between actual and target score on test "deviation right line bisection"

CONTACTS AND LOCATIONS:
Overall Officials: Ruet Alexis, PHD, Principal Investigator — HOPITAL RAYMOND POINCARE
Locations (1):
- Hopital Raymond Poincare Mpr, Garches, Garches, France